CLINICAL TRIAL: NCT02130011
Title: Managing the Real Dose: Evaluating the Impact on Gastric Filling on the Delivered Radiation Dose in Gastrooesophageal Junction Tumors
Brief Title: Dose-Guided Radiotherapy in Oesophageal Cancer: Managing the Real Dose
Acronym: DGRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DGRT; 14-01-15/01-intern-6505 (Other: IRB Maastro Clinic)
Record Dates: First submitted 2014-03-13; First posted 2014-05-02 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- without feeding/fluid instructicon (No Intervention): Ten patients treated with preoperative chemoradiotherapy without feeding/fluid instructions
- with feeding/fluid instructions (Experimental): Ten patients treated with preoperative chemoradiotherapy with feeding/fluid instructions
  Interventions: Other: with feeding/fluid instruction

INTERVENTIONS:
Other: with feeding/fluid instruction — No additional intervention besides standard treatment prescription will be added. Investigators foresee daily kV cone beam CT matching (already standard in house). this subgroup of 10 patients will be asked not to eat or drink carbonated fluids three hours before CT simulation and daily treatment
  Arms: with feeding/fluid instructions

SUMMARY:
This study will prospectively collect patients undergoing the standard CROSS regimen in the neoadjuvant setting of the treatment for gastro-oesophageal cancer. The investigators will focus on the potential geometric differences between the OAR and target volume on the initial planning CT and on the kilovolt (kV) cone-beam computed tomography (CBCT). They expect a potential difference in the abdominal part of the planned target volume (PTV) and/or gastro-oesophageal junction part. Furthermore, the impact of gastric filling , potential tumor regression and the accuracy of 5 mm PTV margin in the thoracic PTV will be monitored.

DETAILED DESCRIPTION:
Optimal radiotherapy planning and delivery is essential for irradiation of gastro-oesophageal junction tumors. There is a need for individualized radiotherapy delivery to the upper abdomen, because of mobility. Likewise, controlling gastric filling by instructing patients about fluid and food intake before treatment, may contribute to positional reproducibility. There is evidence that missing microscopic disease in treating the clinical target volume (CTV) results in a worse prognostic outcome. The investigators want to evaluate wether positional difference of stomach, with and without fasting prescription, has an impact of the delivered dose. They will focus on the part of the CTV extending in the stomach. The investigators hypothesize that measurement of the dose using verification kilovoltage cone beam CTs will provide information on potential cold/hot spots of dose delivery and monitor potential geometric differences during treatment. This may result in a suboptimal treatment and a reconsideration of matching target volume on soft tissue instead of bony landmarks. The investigators will evaluate the first clinical results with DGRT in patients with esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the gastro-oesophageal junction
* Age 18 years or older
* International Union Against Cancer (UICC) T2-4 N0-2 M0, potentially resectable disease treated by the CROSS regimen
* WHO 0-2

Exclusion Criteria:

* Thoracic adenocarcinoma/squamous cell carcinoma
* Palliative treatment for the oesophageal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in which the CTV was not covered | Weekly during radio-and chemotherapy (5 weeks)
  Proportion of patients in which the CTV was not covered (CTV D99, V95, Dmean) with and without different filling status of the stomach in patients treated with neoadjuvant chemoradiotherapy for gastroesophageal cancer

SECONDARY OUTCOMES:
Thoracic margin evaluation | weekly during radio-and chemotherapy (5weeks)
  evaluation if a CTV-PTV margin of 5 mm in the thoracic part of the target volume is sufficient
Stomach variation | Weekly during radio-and chemotherapy (5 weeks)
  stomach movement evaluation on a weekly cone beam CT during chemo radiotherapy with and without feeding/fluid instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, MD, PhD, Principal Investigator — Maastricht Radiation Oncology
Locations (1):
- MAASTRO clinic, Maastricht, Netherlands